CLINICAL TRIAL: NCT06825286
Title: The Effect of Dexmedetomidine as an Adjuvant to Bupivacaine in Ultrasound-Guided Quadratus Lumborum Block for Postoperative Analgesia in Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Dexmedetomidine as an Adjuvant to Bupivacaine in Ultrasound-Guided Quadratus Lumborum Block for Postoperative Analgesia in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Waleed Nagah El said, Resident of Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine,Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS296/8/23
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Dexmedetomidine; Bupivacaine; Ultrasound-Guided; Quadratus Lumborum Block; Postoperative Analgesia; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Bupivacaine; Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine group (Active Comparator): Patients received general anesthesia and bilateral ultrasound guided transmuscular quadratus lumborum block with (20 ml bupivacaine 0.25%)
  Interventions: Drug: Bupivacaine
- Bupivacaine and Dexmedetomidinc group (Experimental): Patients received general anesthesia and bilateral ultrasound guided transmuscular quadratus lumborum block with (20ml Bupivacaine 0.25%) + (Dexmedetomidine I mic/kg)
  Interventions: Drug: Bupivacaine and Dexmedetomidinc) group

INTERVENTIONS:
Drug: Bupivacaine — Patients received general anesthesia and bilateral ultrasound guided transmuscular quadratus lumborum block wilh (20 ml bupivacaine 0.25%).
  Arms: Bupivacaine group
Drug: Bupivacaine and Dexmedetomidinc) group — Patients received general anesthesia and bilateral ultrasound guided transmuscular quadratus lumborum block with (20ml Bupivacaine 0.25%) + (Dexmedetomidine Imic/kg)
  Arms: Bupivacaine and Dexmedetomidinc group

SUMMARY:
The aim of this study is to evaluate the effect of adding Dexmedctomidinc as adjuvant to Bubivacaine in Ultrasound-Guided Quadratus Lumborum Block for Postoperative Analgesia in Laparoscopic Cholecystectomy.

DETAILED DESCRIPTION:
When compared to conventional surgery, laparoscopic cholecystectomy is less invasive and leads to less postoperative pain. However, the postoperative pain following laparoscopic cholecystectomy consists of both somatic and visceral components with pain originating from port entry' wounds, gallbladder resection and abdominal insufflation that leads to peritoneal distention and peritoneal damage.

Quadratus lamborum block (QLB) is abdominal truncal block that provides both somatic and visceral analgesia for both upper and lower abdominal surgical procedures, It was first introduced by Blanco.Currently There are 4 approaches described for QLB: lateral, posterior, anterior and intramuscular. Transmuscular (anterior) QLB Type 3 block involves injection in the plane between the psoas major (PM) and the QL muscles studies have reported spread of the injectate to the thoracic paravertebral space, as well as the spinal nerve which runs anterior to the QL muscle

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-65 years.
* Both genders.
* American society of Anesthesiology (ASA) class l, II undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patient refusal
* History of allergy to local anesthetic.
* Liver or renal pathology affecting drug elimination
* Menta!dysfunction or cognitive disorders.
* Patients on chronic pain medications.
* Body Mass Index > 40 kg/m2.
* Coagulopathy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Intravenous morphine 2 mg given when numerical rating scale equal or above 4 as rescue analgesia

SECONDARY OUTCOMES:
Mean arterial blood pressure | At the end of the operation(Up to 48 min).
  Mean arterial blood pressure was recorded before the block (base-line value), after skin incision by 5,15,30 minutes, and at the end of the operation.
Heart rate | At the end of the operation (Up to 48 min).
  Heart rate was recorded before the block (base-line value), after skin incision by 5,15,30 minutes, and at the end of the operation.
lntraoperative fentanyl consumption | lntraoperatively
  Additional fentanyl dosages of 0.5 µg/kg IV was administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Degree of pain score | 24 hours postoperatively
  Postoperative pain was assessed by the numerical rating scale (NRS; 0 no pain while 10 is the maximum pain) immediately after discharge to the PACU and ward at 6, 12, 18, 24 hours.
Time to the first request for the rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).IV morphine 2mg was given when NRS equal or above 4.
Incidence of Complication | 24 hours postoperatively
  Complication such as bradycardia, hypotension, nausea, vomiting, Pruritis, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author.